CLINICAL TRIAL: NCT06133400
Title: Mapping the Health Status of the Population of French Polynesia: the MATAEA Project
Acronym: MATAEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Louis Malardé (Other)
Collaborators: Institut Pasteur (Industry); Institut de la Statistique de la Polynésie française (Unknown); Centre Hospitalier de la Polynésie française (Unknown); Université de la Polynésie française (Unknown); Institut National en Santé Publique du Québec (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-ILM-001; 2019-A01793-54 (Other: ANSM); 2017-069 (Other: Institut Pasteur)
Record Dates: First submitted 2023-10-30; First posted 2023-11-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Non Communicable Diseases; Microbiome; Communicable Diseases; Pesticide Exposure; Metal Poison; Genetics Population; Ciguatera
Keywords: cross-sectional survey; non-communicable disease; communicable disease; French Polynesia; population genetics
MeSH Terms: conditions — Noncommunicable Diseases; Communicable Diseases; Heavy Metal Poisoning; Ciguatera Poisoning | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects representative of the adult population (18-69 y) of French Polynesia (Experimental): Population sample composed of people aged 18 to 69. These people must have been living in French Polynesia for more than two years at the time of the 2017 census
  Interventions: Other: Questionnaire; Other: Physical measurements; Other: Biological samples

INTERVENTIONS:
Other: Questionnaire — Questionnaire about socio-demographical status, health status and lifestyle habits
Other: Physical measurements — Measurement of height, weight, waist circumference, blood pressure and skin pigmentation
Other: Biological samples — Collect venous blood, saliva and stool samples

SUMMARY:
This is a cross-sectional study carried out on a sample of the adult population aged 18 to 69, distributed over the five archipelagos of French Polynesia.

Participation in the study involves: agreement to answer a questionnaire to collect information on socio-demographic characteristics, lifestyle habits and medical history; physical measurements (height, weight, waist circumference, blood pressure and skin pigmentation); and agreement to take biological samples (blood, saliva and stool) for biological, genetic and microbiological analyses.

The aim of the study is to assess the current health status of the population of French Polynesia and to evaluate the influence of contextual risk factors (lifestyle, place of residence, history of infection) and intrinsic susceptibility factors (genetics, age, gender, microbiota) in relation to non-communicable and infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18 or over and under 70 on the date of recruitment
* having signed the consent form

Exclusion Criteria:

* Minors
* Pregnant or parturient women, and nursing mothers
* Persons deprived of their liberty by a judicial or administrative decision
* Adults who are the subject of a legal protection measure or who are unable to express their consent
* People undergoing psychiatric care
* Individuals who are not affiliated to a social security scheme or beneficiaries of such a scheme
* Homeless people
* Disabled people (unable to move)
* People unable to answer the questionnaire

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1942 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of obesity | 2 years
  Proportion of participants with indicators of obesity based on physical measurements (BMI, waist circumference) and quantification of lipid levels from blood samples.
Prevalence of diabetes | 2 years
  Proportion of participants with indicators of diabetes based on self-reported data on diabetes history (previous diagnosis, antidiabetic treatment) and quantification of glycated haemoglobin from blood samples.
Prevalence of cardiovascular diseases | 2 years
  Proportion of participants with indicators of cardiovascular diseases based on self-reported data on history of hypertension (previous diagnosis, treatment for hypertension), blood pressure measurement, and quantification of lipid levels from blood samples.
Association between non-communicable diseases and behavioral factors | 2 years
  Calculation of odd ratios to investigate association between non-communicable diseases (obesity, diabetes, cardiovascular diseases) and behavioral factors such as tobacco smoking, alcohol consumption, diet or physical activity data self-reported by the participants in the questionnaire.
Association between non-communicable diseases and physical measurements | 2 years
  Calculation of odd ratios to investigate association between non-communicable diseases (obesity, diabetes, cardiovascular diseases) and physical measurements such as BMI (based on the BMI formula i.e., weight in kilograms divided by height in meters squared).
Association between non-communicable diseases and blood analyses | 2 years
  Calculation of odd ratios to investigate association between non-communicable diseases (obesity, diabetes, cardiovascular diseases) and blood analyses (such as glycated haemoglobin and lipid levels).
Seroprevalence of communicable diseases | 2 years
  Proportion of participants with IgG antibodies, detected in blood samples, specific for different pathogens : arboviruses (four dengue serotypes, Zika, chikungunya), hepatitis B and C viruses, hantaviruses, SARS-CoV-2 and other pathogens known to regularly cause infections in French Polynesia (including influenza viruses, human immunodeficiency virus…). Proportion of participants with positive filarial antigenemia to assess the prevalence of Bancroftian lymphatic filariasis.
Composition of microbiome | 2 years
  Bacterial DNA sequencing from stool and saliva samples to assess the gut and oral microbiota profiles and association with lifestyle behavior, diet and susceptibility to communicable and non-communicable diseases.
Level of exposure to heavy metals | 2 years
  Quantification of levels of heavy metals (including mercury and lead) from blood samples and association with lifestyle behavior and diet.
Level of exposure to pesticides | 2 years
  Quantification of levels of pesticides (including chlordane and toxaphene) from blood samples and association with lifestyle behavior and diet.
Level of exposure to mosquito bites | 2 years
  Proportion of participants with IgG antibodies targeting mosquito salivary proteins in blood samples to assess the risk of infection by mosquito-borne viruses
Prevalence of ciguatera poisoning | 2 years
  Estimation of the rate of ciguatera poisoning in the population based on data self-reported by the participants in the questionnaire e.g. the occurrence of symptoms suggestive for ciguatera poisoning at least once in their lifetime
Demographic and adaptive history of French Polynesians using genomics | 2 years
  Human Whole Genome Sequencing from saliva samples to reconstruct the genetic history of the population of French Polynesia, in terms of both demographic and adaptive history.
Genetic susceptibility to obesity | 2 years
  Genome-wide association studies to identify human genetic factors that are associated with BMI or lipids levels.
Genetic susceptibility to diabetes | 2 years
  Genome-wide association studies to identify human genetic factors that are associated with HbA1c.
Genetic susceptibility to communicable diseases | 2 years
  Genome-wide association studies to identify human genetic factors that are associated with the detection of IgG antibodies specific for different pathogens: arboviruses, hepatitis B and C viruses, hantaviruses, SARS-CoV-2 and other pathogens known to regularly cause infections in French Polynesia (including influenza viruses, human immunodeficiency virus…).

CONTACTS AND LOCATIONS:
Overall Officials: Van-Mai CAO-LORMEAU, PhD, Study Director — Institut Louis Malardé
Locations (1):
- Institut Louis Malardé, Papeete, Îles du Vent, French Polynesia

REFERENCES:
- [Derived] Teiti I, Aubry M, Fernandes-Pellerin S, Patin E, Madec Y, Boucheron P, Vanhomwegen J, Torterat J, Lastere S, Olivier S, Jaquaniello A, Roux M, Mendiboure V, Harmant C, Bisiaux A, Rijo de Leon G, Liu D, Bossin H, Mathieu-Daude F, Gatti C, Suhas E, Chung K, Condat B, Ayotte P, Conte E, Jolly N, Manuguerra JC, Sakuntabhai A, Fontanet A, Quintana-Murci L, Cao-Lormeau VM. Unravelling the determinants of human health in French Polynesia: the MATAEA project. Front Epidemiol. 2023 Nov 27;3:1201038. doi: 10.3389/fepid.2023.1201038. eCollection 2023. PMID 38455935